CLINICAL TRIAL: NCT02046746
Title: The Effect of a Renal Specific Oral Nutritional Supplement on Nutritional Status and Other Outcomes
Brief Title: The Effect of a Renal Specific Oral Nutritional Supplement on Nutritional Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DA03
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral Nutritional Supplement (ONS) (Experimental): 1-2 serving per day of a renal specific oral nutritional supplement
  Interventions: Other: Oral Nutritional Supplement (ONS)

INTERVENTIONS:
Other: Oral Nutritional Supplement (ONS) — renal specific commercially available ONS

SUMMARY:
The study objective is to evaluate if a renal specific oral nutrition supplement (ONS) aids in maintaining nutritional status.

DETAILED DESCRIPTION:
This study is an unblinded, prospective, multicenter, single arm study in Taiwan. Eligible subjects (see inclusion and exclusion criteria in Section 5.2) will receive standard of care (which includes dietary counseling) and ONS supplementation (1-2 servings/day depending on subject's needs) for 24 weeks (6 months). A follow up visit (phone call/medical chart review) will occur 12 months after the study intervention has ended to collect mortality data, to determine whether or not dialysis was initiated, and if ONS use continued.

Subjects will be informed of the study results when available. Subjects may continue use of the commercially available study product if it is recommended by their nephrologist, primary care physician, dietitian, or if the subject chooses.

For this study enrollment is defined as when the subject is stratified and begins to consume the study product (Study Visit 1, Month 0).

The target population described above may be stratified into the following groups (n=18 evaluable/group):

1. Male CKD Stage 3b-5 without T2DM
2. Male CKD Stage 3b-5 with T2DM
3. Female CKD Stage 3b-5 without T2DM
4. Female CKD Stage 3b-5 with T2DM

In addition, for those subjects enrolled, retrospective data (previous 6 to 12 months) identical to the study variables will be collected. Retrospective data collection will focus on the following measures, however, all data points are not expected to be available:

* Serum albumin
* SGA
* Compliance to protein intake guidelines
* Compliance to energy intake guidelines
* Hand grip strength
* Anthropometrics (weight, height, BMI)
* Quality of Life (WHOQOL-BREF Taiwan Version)
* eGFR (whichever equation is used as standard of care)
* Serum creatinine
* Proteinuria (retrospective - if available on medical records)
* BUN
* Body composition data from BIA (especially fat mass and muscle mass, units or exact terminology will be model specific)
* C reactive protein (CRP)
* Blood chemistries,

ELIGIBILITY:
Inclusion Criteria:

1. Subject, or subject's legally acceptable representative (LAR), has voluntarily signed and dated an informed consent form (ICF), approved by an IEC/IRB, and provided Health Insurance Portability and Accountability Act (HIPAA)
2. Subject is >18 years of age.
3. Subject has been diagnosed with Chronic Kidney Disease (CKD) and is classified as being between Stages 3b to 5.
4. Subject has an eGFR 45 and 10 ml/min/1.73m2 at screening.
5. Subject is a male or non-pregnant female at least six weeks postpartum and non-lactating.
6. Subject with CKD is either:

   * not diagnosed with Type 2 Diabetes Mellitus (T2DM) OR
   * diagnosed with T2DM and had no changes in glycemic medication (dose or type) for at least 2 months prior to screening
7. Subject has a serum albumin 3.0 g/dl at screening.
8. Subject has a BMI 30 kg/m2.
9. If diagnosed with T2DM, subject has A1c level 9.0% at screening.
10. Subject is not scheduled or expected to receive dialysis in the next 18 months.
11. Subject's life expectancy is 18 months determined by the study physician.
12. Subject is willing to follow the protocol as described.
13. With regard to ONS use the subject must qualify as one of the following:

    1. be naïve to ONS
    2. if the subject is already prescribed another ONS that is not the study product, and they have consumed 8 servings over the last 28 days prior to screening, they will undergo a washout period (3 weeks)
    3. if the subject is already prescribed the study product, and they have consumed ≤ 8 servings over the last 28 days prior to screening, or have poor daily compliance (< 75%), they will undergo a washout period (3 weeks)
    4. if the subject is already prescribed the study product, and they have been consuming 1-2 servings daily, with >75% compliance, for < 3 months, they do not require a washout period, and can be retrospectively included in the study protocol (provided proper records can be obtained)

Exclusion Criteria:

1. Subject has type 1 diabetes.
2. Subject is considered malnourished (SGA = 1 to 3).
3. Subject has received intravenous albumin treatment within the last 6 months.
4. Subject has overt symptomatic peripheral neuropathy, retinopathy, or autonomic neuropathy.
5. Subject has poorly controlled chronic hypertension
6. Subject has had major surgery, inpatient or outpatient, requiring >7 days of hospitalization in the last 3 weeks prior to screening visit,
7. Subject has a known chronic/contagious infectious disease, clotting or bleeding disorder, active malignancy
8. Subject is missing, or has had an amputation of, a limb.
9. Subject has had a significant cardiovascular event
10. Subject has a known obstruction of the gastrointestinal tract, inflammatory bowel disease, short bowel syndrome or other forms of gastrointestinal disease
11. Subject is currently diagnosed with, or has a history of severe dementia or delirium, eating disorder, history of significant neurological or psychiatric disorder, alcoholism, substance abuse or other conditions that may interfere with study product consumption or compliance with study protocol procedures
12. Subject is currently consuming, or cannot refrain from taking, medications/dietary supplements/herbal preparations or substances,
13. Subject is known to be allergic or intolerant to any ingredient found in the study product.
14. Subject is considered unsuitable for the study based on the study physician's assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-11; Primary Completion 2016-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Serum Albumin | Change from Month 0 to Month 6

SECONDARY OUTCOMES:
Subjective Global Assessment | Change from Month 0 to Month 6
Dietary Intake Compliance | Change from Month 0 to Month 6
Hand Grip Strength | Change from Month 0 to Month 6
Appetite | Change from Month 0 to Month 6
Body Mass Index | Change from Month 0 to Month 6
Quality of Life | Change from Month 0 to Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Owen Kelly, Ph.D, Study Chair — Abbott Nutrition
Locations (2):
- Taiwan (2):
  - Kaohsiung Medical University Hospital (KMUH), Kaohsiung City
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No